CLINICAL TRIAL: NCT00281957
Title: A Randomized Phase II Trial of BAY 43-9006 (Sorafenib; NSC-724772) With Either CCI-779 (Temsirolimus; NSC-683864) or R115777 (Tipifarnib; NSC-702818) in Metastatic Melanoma
Brief Title: Sorafenib With Either Temsirolimus or Tipifarnib in Treating Patients With Stage IV Malignant Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00774; NCI-2009-00774 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0438; CDR0000454925; S0438 (Other: SWOG); S0438 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; tipifarnib; temsirolimus; Sirolimus

ARMS (2):
- Arm I (sorafenib, temsirolimus) (Experimental): Patients receive oral sorafenib twice daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: sorafenib tosylate; Drug: temsirolimus
- Arm II (sorafenib, tipifarnib) (Experimental): Patients receive oral sorafenib as in arm I and oral tipifarnib twice daily on days 1-21
  Interventions: Drug: sorafenib tosylate; Drug: tipifarnib

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
  Arms: Arm II (sorafenib, tipifarnib)
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
  Arms: Arm I (sorafenib, temsirolimus)

SUMMARY:
This randomized phase II trial is studying how well giving sorafenib together with either temsirolimus or tipifarnib works in treating patients with stage IV melanoma that cannot be removed by surgery. Sorafenib, temsirolimus, and tipifarnib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib and tipifarnib may also stop the growth of tumor by blocking blood flow to the tumor. It is not yet known whether sorafenib is more effective when given together with temsirolimus or tipifarnib in treating patients with malignant melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the response rate (confirmed and unconfirmed and complete and partial) in patients with unresectable stage IV malignant melanoma treated with sorafenib in combination with either temsirolimus or tipifarnib.

II. Compare the 4-month progression-free survival rate of patients treated with these regimens.

III. Compare the safety and tolerability of these regimens, with an emphasis on long-term side effects and toxic effects, in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to metastatic (M) stage (M1a/b vs M1c). Patients are randomized to 1 of 2 treatment arms.

ARM I (reopened to accrual as of 8/15/2009): Patients receive oral sorafenib twice daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.

ARM II (closed to accrual as of 8/15/2009): Patients receive oral sorafenib as in arm I and oral tipifarnib twice daily on days 1-21.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Criteria:

* Histologically confirmed malignant melanoma of cutaneous origin
* Patients with unknown primary allowed
* Stage IV disease
* Measurable disease by physical examination, CT scan, MRI or plain x-ray
* Unresectable disease
* Residual or recurrent disease after prior surgery for stage IV disease allowed
* Residual tumor at the site of incomplete resection may be included only as nonmeasurable disease
* Must have serum lactate dehydrogenase (LDH) levels measured
* Must have tissue specimens available
* Negative brain CT scan or MRI within the past 42 days
* Creatinine =< 1.5 times ULN
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Fasting cholesterol =< 350 mg/dL (lipid-lowering agents allowed)
* Triglycerides =< 300 mg/dL (lipid-lowering agents allowed)
* No symptomatic sensory neuropathy >= grade 2
* No evidence of bleeding diathesis or coagulopathy
* No congestive heart failure
* No myocardial infarction within the past 2 months
* No New York Heart Association class III or IV heart disease
* No condition that impairs the ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication, requirement for IV alimentation, prior surgical procedure affecting absorption, or active peptic ulcer disease)
* No known allergy to imidazoles (e.g. clotrimazole, ketoconazole, miconazole, or econazole)
* No history of allergic reaction to compounds of similar chemical or biologic composition as tipifarnib
* No hypertension with systolic blood pressure (BP) > 140 mm Hg or diastolic BP > 90 mm Hg
* Patients with well-controlled hypertension allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled diabetes
* No uncontrolled diabetes
* No active uncontrolled infection
* No other severe or uncontrolled medical disease
* No psychologic or medical condition that would preclude study treatment or compliance
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, adequately treated stage I or II cancer that is in complete remission, or carcinoma in situ of the cervix
* At least 90 days since prior adjuvant therapy, including cytotoxic agents
* At least 28 days since prior radiotherapy
* At least 28 days since prior surgery to remove the tumor
* No prior systemic therapy for stage IV melanoma
* No prior therapy with agents targeting farnesyl transferase, the MAP kinase pathway, or vascular endothelial growth factors (VEGF) or receptors (VEFGR), including drugs such as sorafenib, temsirolimus, or tipifarnib
* Concurrent lipid-lowering agents allowed
* Not requiring full-dose anticoagulation for recent thrombotic event
* No concurrent highly active antiretroviral therapy (HAART) in HIV-positive patients
* No concurrent use of any of the following: dilantin; carbamazepine; Phenobarbital; rifampin; hypericum perforatum (St. John's wort); ketoconazole; itraconazole; ritonavir; cyclosporine; phenytoin; grapefruit juice
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* SGOT or SGPT =< 2.5 times ULN (5 times ULN if hepatic metastases)
* No history of brain metastases
* Zubrod performance status 0-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Margolin, Principal Investigator — SWOG Cancer Research Network
Locations (173):
- United States (173):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Orange Regional Medical Center, Middletown, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Mansfield General Hospital-MedCentral Health System, Mansfield, Ohio
  - Adventist Medical Center, Portland, Oregon
  - SWOG, Portland, Oregon
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib + Temsirolimus: Patients receive oral sorafenib twice daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
- Sorafenib + Tipifarnib: Patients receive oral sorafenib as in arm I and oral tipifarnib twice daily on days 1-21
Period: Overall Study
Arm/Group | Sorafenib + Temsirolimus | Sorafenib + Tipifarnib
Started | 67 | 42
Eligible | 66 | 40
Eligible and Received Treatment | 63 | 39
Completed | 0 | 0
Not Completed | 67 | 42
Not completed — Adverse Event | 7 | 2
Not completed — Death | 1 | 0
Not completed — Progression/relapse | 47 | 35
Not completed — Not protocol specified | 8 | 1
Not completed — Not eligible | 1 | 2
Not completed — Did not start treatment | 3 | 1
Not completed — Refusal unrelated to adverse events | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Sorafenib + Temsirolimus: Patients receive oral sorafenib twice daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
- Arm II: Sorafenib + Tipifarnib: Patients receive oral sorafenib as in arm I and oral tipifarnib twice daily on days 1-21
- Total: Total of all reporting groups
Arm/Group | Arm I: Sorafenib + Temsirolimus | Arm II: Sorafenib + Tipifarnib | Total
Number analyzed (Participants) | 63 | 39 | 102
Age, Continuous [Median (Full Range); unit: years] | 64 [27 to 85] | 58 [28 to 84] | 62 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 17 | 46
  Male | 34 | 22 | 56
Region of Enrollment [Number; unit: participants]
  United States | 63 | 39 | 102

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial)
Description: Complete response corresponds to complete disappearance of all measurable and non-measurable lesions with no new lesions. Partial response corresponds to greater than or equal to 30ﬁ decrease of sum of longest diameter of all target measurable lesions with no new lesion and non unequivocal progression of non-measurable disease.
Time Frame: Every 8 weeks until progression
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Sorafenib+Temsirolimus: Patients receive oral sorafenib twice daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
- Sorafenib+Tipifarnib: Patients receive oral sorafenib as in arm I and oral tipifarnib twice daily on days 1-21
Arm/Group | Sorafenib+Temsirolimus | Sorafenib+Tipifarnib
Number analyzed (Participants) | 63 | 39
Percent of participants | 5 [1 to 13] | 3 [0 to 13]

2. Primary Outcome: 4-month Progression-free Survival
Description: Progression was defined as one or more of the following: 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed, unequivocal progression of non-measurable disease, appearance of any new lesions, death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: 4 months after registration
Measure: Number (95% Confidence Interval); unit: Percent of population
Arm/Group | Sorafenib+Temsirolimus | Sorafenib+Tipifarnib
Number analyzed (Participants) | 63 | 39
Percent of population | 29 [19 to 41] | 18 [8 to 31]

3. Secondary Outcome: One-year Overall Survival
Time Frame: One year after registration
Measure: Number (95% Confidence Interval); unit: Percent of population
Arm/Group | Sorafenib+Temsirolimus | Sorafenib+Tipifarnib
Number analyzed (Participants) | 63 | 39
Percent of population | 19 [11 to 30] | 31 [17 to 45]

4. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: Weekly during first cycle, every two weeks during the second cycle, and once a cycle further cycles (one cycle = 4 weeks).
Population: Eligible patients who had received any hydroxyurea
Measure: Number; unit: Participants
Groups:
- Sorafenib+Temsirolimus: Sorafenib and Temsirolimus
- Sorafenib+Tipifarnib: Sorafenib and Tipifarnib
Arm/Group | Sorafenib+Temsirolimus | Sorafenib+Tipifarnib
Number analyzed (Participants) | 63 | 39
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 1
  AST, SGOT (serum glut oxaloacetic transaminase) | 0 | 1
  Amylase | 0 | 1
  Anorexia | 1 | 0
  Calcium, serum-low (hypocalcemia) | 1 | 0
  Confusion | 2 | 0
  Constitutional Symptoms-Other (Specify) | 1 | 0
  Cough | 1 | 0
  Creatinine | 1 | 0
  Dehydration | 3 | 0
  Dermatology/Skin-Other (Specify) | 0 | 1
  Diarrhea | 4 | 1
  Dyspnea (shortness of breath) | 1 | 1
  Fatigue (asthenia, lethargy, malaise) | 8 | 2
  Gastrointestinal-Other (Specify) | 1 | 0
  Glucose, serum-high (hyperglycemia) | 1 | 0
  Heartburn/dyspepsia | 0 | 1
  Hemoglobin | 2 | 0
  Hemorrhage, GI - Stomach | 1 | 0
  Hypertension | 1 | 2
  Hypotension | 1 | 0
  Ileus, GI | 1 | 0
  Infec with norm ANC or Gr 1/2 neut- Nose | 1 | 0
  Infec with norm ANC or Gr 1/2 neut-Skin | 1 | 0
  Left ventricular systolic dysfunction | 1 | 0
  Lipase | 0 | 1
  Lymphopenia | 1 | 0
  Mood alteration - depression | 0 | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2 | 0
  Muscle weakness, gen or spec area-Extraocular | 1 | 0
  Muscle weakness, gen or spec area-Whole body | 2 | 1
  Nausea | 3 | 0
  Neurology-Other (Specify) | 1 | 0
  Neuropathy: motor | 0 | 1
  Obstruction, GI - Small bowel NOS | 1 | 0
  Pain - Abdomen NOS | 1 | 2
  Pain - Back | 1 | 2
  Pain - Chest wall | 1 | 0
  Pain - Chest/thorax NOS | 1 | 1
  Pain - Extremity-limb | 1 | 1
  Pain - Head/headache | 1 | 0
  Pain - Joint | 1 | 1
  Pain - Muscle | 1 | 0
  Pain - Neuralgia/peripheral nerve | 0 | 1
  Pain - Oral cavity | 1 | 0
  Pain - Pelvis | 0 | 1
  Pain - Rectum | 1 | 0
  Pain - Skin | 1 | 0
  Pain - Stomach | 1 | 0
  Pancreatitis | 1 | 1
  Phosphate, serum-low (hypophosphatemia) | 8 | 1
  Platelets | 1 | 0
  Pneumonitis/pulmonary infiltrates | 2 | 0
  Potassium, serum-low (hypokalemia) | 4 | 0
  Proteinuria | 1 | 0
  Pruritus/itching | 2 | 1
  Pulmonary/Upper Respiratory-Other (Specify) | 1 | 0
  Rash/desquamation | 4 | 2
  Rash: acne/acneiform | 3 | 5
  Rash: erythema multiforme | 1 | 0
  Rash: hand-foot skin reaction | 2 | 4
  Renal failure | 2 | 0
  Sodium, serum-low (hyponatremia) | 1 | 0
  Thrombosis/thrombus/embolism | 0 | 1
  Vomiting | 3 | 0

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Groups:
- Arm I: Sorafenib and Temsirolimu
- Arm II: Sorafenib and Tipifarnib
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 13/63 | 6/39
Other Adverse Events (participants affected / at risk) | 61/63 | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=63) | Arm II (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Nose (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 | 0
Amylase (Investigations) | 0 | 1
Lipase (Investigations) | 0 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 0
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Neurology-Other (Specify) (Nervous system disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 1
Pain - Head/headache (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=63) | Arm II (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 28 | 3
Constipation (Gastrointestinal disorders) | 7 | 8
Diarrhea (Gastrointestinal disorders) | 18 | 17
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 13 | 4
Nausea (Gastrointestinal disorders) | 21 | 7
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 9 | 2
Edema: limb (General disorders) | 5 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 42 | 22
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 7 | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 14 | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 15 | 2
Alkaline phosphatase (Investigations) | 9 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 2
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 25 | 7
Creatinine (Investigations) | 9 | 2
Leukocytes (total WBC) (Investigations) | 15 | 0
Lymphopenia (Investigations) | 5 | 0
Metabolic/Laboratory-Other (Specify) (Investigations) | 8 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 | 0
Platelets (Investigations) | 20 | 3
Weight loss (Investigations) | 13 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9 | 4
Anorexia (Metabolism and nutrition disorders) | 20 | 9
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 14 | 4
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 18 | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 | 3
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 23 | 8
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 2
Neuropathy: sensory (Nervous system disorders) | 5 | 6
Pain - Head/headache (Nervous system disorders) | 7 | 3
Taste alteration (dysgeusia) (Nervous system disorders) | 11 | 0
Insomnia (Psychiatric disorders) | 4 | 2
Mood alteration - depression (Psychiatric disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 6
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 | 9
Rash/desquamation (Skin and subcutaneous tissue disorders) | 18 | 11
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 21 | 13
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5 | 7
Flushing (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less